CLINICAL TRIAL: NCT00676884
Title: A Phase 2a Study to Investigate the Effects of Repeated Administration of AeroDerm in Subjects With Atopic Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerovance, Inc. (Industry)
Responsible Party: Rick Fuller, FRCP, Aerovance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QGUY/2005/AER 001/-02
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Atopic Eczema
Keywords: atopic eczema; atopic dermatitis; allergy
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity | interventions — pitrakinra; 5-methoxy-methylindoleacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aeroderm (also known as pitrakinra, AER 001, BAY 16-9996)
  Interventions: Drug: Aeroderm (also known as pitrakinra, AER 001, BAY 16-9996)
- 2 (Placebo Comparator): placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aeroderm (also known as pitrakinra, AER 001, BAY 16-9996) — 30 mgs s.c. b.i.d.
  Other Names: AER 001, BAY16-9996, pitrakinra
  Arms: 1
Drug: placebo — 1.5 mL s.c. b.i.d.
  Other Names: pbs
  Arms: 2

SUMMARY:
The primary objective of this study is to investigate the effect of AERODERM (also known as pitrakinra, AER 001, BAY 16-9996) on Eczema Area and Severity Index (EASI) score in subjects with moderate to severe atopic eczema

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the effect of AERODERM (also known as pitrakinra, AER 001, BAY 16-9996) on Eczema Area and Severity Index (EASI) score in subjects with moderate to severe atopic eczema in a randomised, placebo controlled, parallel-group study with bid sc. dosing of AERODERM for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females > 18 years.
* Subjects who currently have allergic eczema with an EASI score in the range of 10-50.
* Subjects who have been on a stable dose of topical medications for eczema for ≥ 1 month from screening but whose eczema is not adequately responsive to, or controlled by, conventional topical treatments (eg: topical steroids, Tracrolimus, Pimecrolimus).
* Subjects who have not had systemic immunosuppressive therapy (eg systemic steroids) within 1 month of screening.
* Subjects who if female, are not currently pregnant or breast feeding and are using medically acceptable methods of contraception.
* Subjects who have a pre-study medical history, physical examination and vital signs acceptable to the investigator.
* Subjects who have clinical laboratory tests within the reference ranges or clinically acceptable to the investigator.
* Subjects who are negative for HbsAg, hepatitis C antibody and HIV II and I test at screening.
* Subjects who are negative for drugs of abuse tests at screening and admission.
* Subjects with stable, adequately treated medical conditions other than eczema may be enrolled provided the Investigator does not consider their study participation to place them at increased risk of adverse events. Subjects should continue their concomitant treatments for medical conditions (other than eczema).
* Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who do not conform to the above inclusion criteria.
* Subjects who have the following medical conditions: Diabetes mellitus, Thyroiditis, Rheumatiod arthritis, Multiple sclerosis, Uveitis, Sarcoidosis, Glomerulonephritis, Helminthic infection.
* Subjects who have a history of relevant drug hypersensitivity.
* Subjects who have a history of alcoholism.
* Subjects who have a history of drug abuse.
* Subjects who have a significant infection at the time of screening and/or admission.
* Subjects who are having acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn), may be asked to reschedule their screening and/or admission to when they are not longer having acute symptoms.
* Subjects who have an acute infection such as influenza at the time of screening and/or admission.
* Female subjects who are not using an acceptable method of contraception.
* Subjects who have used any investigational drug and /or participated in any clinical trial within 3 months of their first dosing.
* Subjects who have previously received AeroDerm.
* Subjects using medication, which in the opinion of the Investigator will affect the outcome of the study.
* Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to first dosing (to review on a case by case basis).
* Subjects who cannot communicate reliably with the investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity index (EASI) score | weekly for 28 days of treatment

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) | daily for 28 days of treatment
levels of Tcell subsets | after 28 days of treatment
total IgE | after 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, Principal Investigator — Guy's Drug Research Unit, Quintiles Limited; Richard Groves, FRCP, Principal Investigator — St. Johns Institute of Dermatology St. Thomas' Hospital London
Locations (1):
- Guy's Drug Research unit, Quintiles Limited, London, United Kingdom